CLINICAL TRIAL: NCT01414556
Title: Effects of Glucose-dependent Insulinotropic Polypeptide at Insulin Induced Hypoglycemia in Patients With Type 2 Diabetes
Brief Title: GIP Effects at Insulin Induced Hypoglycemia in Patients With Type 2 Diabetes
Acronym: GIP-HYPO-T2DM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mikkel Christensen (Other)
Responsible Party: Sponsor-Investigator, Mikkel Christensen, MD, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-2-2009-078
Record Dates: First submitted 2011-08-05; First posted 2011-08-11 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Incretins; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- hyperglycemia (Experimental)
  Interventions: Other: Glucose-dependent Insulinotropic polypeptide; Other: saline
- fasting glycemia (Experimental)
  Interventions: Other: Glucose-dependent Insulinotropic polypeptide; Other: saline
- hypoglycemia (Experimental)
  Interventions: Other: Glucose-dependent Insulinotropic polypeptide; Other: saline

INTERVENTIONS:
Other: Glucose-dependent Insulinotropic polypeptide — infusion 4 pmol x kg x min first 15 min, thereafter 2 pmol x kg x min
Other: saline

SUMMARY:
Investigation of GIP effects at fasting and hypoglycemia

ELIGIBILITY:
Inclusion Criteria:

* Caucasians 18 years or older with Type 2 diabetes (WHO criteria)

Exclusion Criteria:

* HbA1c >9 %
* Liver disease (ALAT/ASAT >2 x upper normal limit)
* Diabetic nephropathy (s-creatinine >130 µM or albuminuria)
* Proliferative diabetic retinopathy (anamnestic)
* Severe arteriosclerosis or heart failure (NYHA group III og IV)
* Anemia
* treatment with medication not applicable to pause for 12 hours
* Fasting plasma glucose >15 mM on screening day.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
glucagon/insulin(c-peptide) absolute, incremental and area under curve values | approx. 15 minutes intervals, time 0 to 120 min

SECONDARY OUTCOMES:
plasma gut hormones and nutrients | approx. 15 minutes intervals, time 0 to 120 min

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte Hospital, Hellerup, Denmark

REFERENCES:
- [Derived] Veedfald S, Vedtofte L, Skov-Jeppesen K, Deacon CF, Hartmann B, Vilsboll T, Knop FK, Christensen MB, Holst JJ. Glucose-Dependent Insulinotropic Polypeptide Is a Pancreatic Polypeptide Secretagogue in Humans. J Clin Endocrinol Metab. 2020 Mar 1;105(3):dgz097. doi: 10.1210/clinem/dgz097. PMID 31665480
- [Derived] Christensen MB, Calanna S, Holst JJ, Vilsboll T, Knop FK. Glucose-dependent insulinotropic polypeptide: blood glucose stabilizing effects in patients with type 2 diabetes. J Clin Endocrinol Metab. 2014 Mar;99(3):E418-26. doi: 10.1210/jc.2013-3644. Epub 2013 Dec 11. PMID 24423311